CLINICAL TRIAL: NCT04491396
Title: Assessing a Gentle Yoga Combined With Yoga Breathing (GYYB) Adjunct Intervention for Scleroderma Self-Management
Brief Title: Yoga Adjunct for Scleroderma
Acronym: GYYB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Richard Silver (Unknown); Marvella Ford (Unknown); Paul Nietert (Unknown); Therese Killeen (Unknown)
Responsible Party: Principal Investigator, Sundaravadivel Balasubramanian, Assistant Professor Research, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12771
Record Dates: First submitted 2020-07-23; First posted 2020-07-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Intervention Model Description: Mixed methods model
Masking Description: The study is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GYYB (Other): This is a single-arm pre-post design.
  Interventions: Behavioral: Gentle Yoga and Yogic Breathing

INTERVENTIONS:
Behavioral: Gentle Yoga and Yogic Breathing — Gentle Yoga (GY) postures can be done while seated on a chair (sometimes called "Chair Yoga") and have been shown to benefit people with symptoms associated with cancer.12 However, Yoga is under-studied in the area of scleroderma. While most traditional Yoga postures can be practiced by anyone, people with scleroderma often have limited physical movement and can be prone to injury. Gentle Yoga postures are physically much easier to do than traditional Yoga and, thus, may be more accessible for SSc patients with musculoskeletal and other impairments. Gentle Yoga postures that are done while seated on a chair also combine easily with YB, but little is known about the specific benefits of the GY+YB combination (GYYB). Further study is needed to determine whether GYYB may be an effective strategy for improving QoL in SSc patients. The Yoga intervention to be used in this study specifically involves GY done while seated in combination with YB.
  Other Names: Chair Yoga and Pranayama

SUMMARY:
This is a pilot research study to determine the feasibility of gentle yoga and breathing exercises for symptom management in patients with scleroderma. Participants will have a first study visit that includes completing demographic and quality-of-life surveys, learning the gentle yoga and breathing exercises, and providing two saliva samples before and after doing the exercises. After this visit, participants will do the gentle yoga and breathing exercises twice daily at home (morning and evening) by following a video hyperlink. Participants will make an entry in their Yoga Practice Diaries each time they practice at home. On the 12th Week, participants will return to MUSC for a final study visit that includes doing the gentle yoga and breathing exercises, providing saliva samples, and completing a satisfaction survey. There will be a total of 2 clinic visits (on Weeks 1 and 12). The study coordinator will telephone participants weekly during the 10 weeks that they do the gentle yoga and breathing exercises at home to answer questions and help solve any problems. Each visit will take about 2 hours for this research study, in addition to any routine clinical examinations. Each home yoga and breathing practice will take 1 hour. The total study duration is 12 Weeks (3 months). Participants will receive compensation for their travel in the form of prepaid Visa gift cards.

DETAILED DESCRIPTION:
This pilot research project will:

* Test the feasibility of a scleroderma self-management intervention that combines Gentle Yoga postures and Yoga Breathing (GYYB) as adjunctive treatment with standard care.
* Explore the effectiveness of GYYB for improving health-related quality-of-life (QoL) outcomes.
* Provide information about acceptance and adoption of a GYYB intervention by scleroderma patients of African ancestry (AA) and non-Hispanic white (NHW) scleroderma patients in the United States (US).
* Investigate, for the first time in scleroderma patients, the relationship between GYYB and inflammatory biomarker changes which may provide insight into biological changes associated with improved health-related QoL outcomes.

The following specific aims will be examined in a Pre/Post design using a 12-week GYYB intervention as an adjunct self-management strategy along with usual care:

Specific Aim 1: Conduct a feasibility trial to assess changes in self-reported QoL in a 12-week adjunct GYYB program among scleroderma patients (N=30) receiving usual care. Outcomes will be assessed in the overall study population and stratified by race/ethnicity (NHW vs. AA).

Specific Aim 2: Assess changes in the expression of inflammatory biomarkers in a 12-week adjunct GYYB program in scleroderma patients receiving usual care. Outcomes will be assessed in the overall study population and stratified by race/ethnicity (NHW vs. AA).

This is a pilot study and will not test a hypothesis. There are no preliminary data for making assumptions regarding effect sizes and variability between Pre/Post measures in this intervention. The main goal of this pilot study is estimation.

Results will provide critical preliminary data for planning a larger study and information about differences (or lack thereof) by race/ethnicity. With N=30 patients overall (n=15 per race/ethnicity group), investigators will be able to obtain relatively precise estimates of completion rates (e.g., 95% confidence intervals extending ±14% for the entire group and extending ±20% for each race/ethnicity group). Assuming some drop-outs over the study (i.e., with n=26 completers), investigators will be able to estimate changes in expression of inflammatory biomarkers with adequate precision (e.g., 95% confidence intervals extending ±0.4 standard deviation units for the entire group and extending ±0.5 standard deviation units for each race/ethnicity group). Although hypothesis testing is secondary, note that this study will have 80% power to detect changes equivalent to 0.6 standard deviation units in the overall sample and 0.8 standard deviation units in each race/ethnicity group (NHW and AA).

ELIGIBILITY:
Inclusion Criteria:

* Men and women fulfilling the 2013 ACR/EULAR Classification for Systemic Sclerosis
* Self-identified race/ethnicity as AA or NHW
* Undergoing treatment from any healthcare provider
* 18 years of age or older
* Ability to perform the study exercises involving gentle movements sitting on a chair and regulated breathing
* Access to a working telephone
* Access to watch a video from a DVD or from a website or Youtube

Exclusion Criteria:

* Diagnosed with psychiatric or cognitive disorder that precludes provision of written informed consent
* Physical limitations making Yoga techniques detrimental
* Enrolled in any other Yoga related clinical trials
* Currently engaged in regular Yoga activity (once per week or more).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Quality of life determination: SHAQ-DI | 12 weeks
  Scleroderma Health Assessment Questionnaire and Disability Index (SHAQ-DI)
Perceived Stress | 12 weeks
  Perceived Stress Scale
Depression | 12 weeks
  10-item Center for Epidemiologic Studies Depression Scale
Salivary biomarkers | Weeks 0 and 12
  IL-1β, IL-8 , IL-6, and MCP-1, and cortisol
Feasibility test | Week 12
  enrollment data
Adherence | 12 weeks
  Practice diary
Acceptance | 12 weeks
  Satisfaction using likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Non-identifiable study results will be shared with the patient and scientific community.